CLINICAL TRIAL: NCT01665690
Title: A Community-level RCT of Expedited Partner Treatment for Gonorrhea and Chlamydia
Brief Title: Washington State Community Expedited Partner Treatment (EPT) Trial
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Washington State, Department of Health (Other Government); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Matthew Golden, Professor, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 29923-J; 5R01AI068107 (NIH)
Record Dates: First submitted 2012-08-13; First posted 2012-08-15 (Estimated); Last update posted 2012-08-17 (Estimated); Status verified 2012-08

CONDITIONS: Gonorrhea; Neisseria Gonorrhoeae; Chlamydia Trachomatis
Keywords: patient delivered partner therapy; expedited partner therapy; partner notification; gonorrhea; chlamydia
MeSH Terms: conditions — Gonorrhea; Chlamydia Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention period (Experimental): The study will include 23 WA state local health jurisdictions (LHJ). Each LHJ will be a randomized unit and a unit in which we will measure outcomes. (LHJs are governmental administrative units that usually correspond with a county.) Because this is a stepped-wedge randomized trial, the study will have two groups (intervention and control). However, each LHJ will be in both groups depending on the time period.
  Interventions: Other: Patient delivered partner therapy; Behavioral: Targeted public health partner services
- Control Period (No Intervention): The study will include 23 WA state local health jurisdictions (LHJ). Each LHJ will be a randomized unit and a unit in which we will measure outcomes. (LHJs are governmental administrative units that usually correspond with a county.) Because this is a stepped-wedge randomized trial, the study will have two groups (intervention and control). However, each LHJ will be in both groups depending on the time period.

INTERVENTIONS:
Other: Patient delivered partner therapy — The study will provide communities with access to free PDPT for heterosexuals with gonorrhea or chlamydial infection. PDPT will be packaged to meet the requirements of the WA State Board of Pharmacy and will include 1gram of azithromycin, information about STD, condoms, and information about enclosed medication in English and Spanish. PDPT packs for gonorrhea will also include 400mg of cefixime.
  Arms: Intervention period
Behavioral: Targeted public health partner services — During intervention periods, communities will receive public health partner services (PS) provided by Disease Intervention Specialists (DIS). Diagnosing clinicians will triage their patients to receive PS based on defined criteria associated with not ensuring partners' treatment. PS will include an offer to notify partners for each index case. When DIS notify partners they will offer them the opportunity to obtain free medication at a local pharmacy, at a clinic (as available) or through the mail. DIS will also offer to refer partners for complete evaluations insofar as such care is available in local communities.
  Arms: Intervention period

SUMMARY:
The Washington State Community Expedited Partner Therapy Trial is a stepped-wedge community level randomized trial designed to test the hypothesis that a public health program designed to increase the use of expedited partner therapy can decrease the prevalence of chlamydial infection in young women and the incidence of gonorrhea in Washington state. The study intervention will be modeled after and intervention previously evaluated in King County WA (Golden MR, Sex Transm Dis 2007;598-603). The intervention has two components: 1) promotion of patient delivered partner therapy (PDPT) use by medical providers in accordance with Washington state guidelines; and 2) targeted provision of partner services. PDPT use will be promoted through education and by making medication packs for PDPT available statewide. Medical providers will refer selected persons with gonorrhea or chlamydial infection for partner services based on defined criteria associated with failure to ensure partners' treatment. The intervention will be instituted in four waves separated by 6-9 months. Each wave will include approximately 6 local health jurisdictions. The order in which health jurisdictions initiate the intervention will be randomly assigned. The study's primary endpoint will be the prevalence of chlamydial infection in women age 15-25 tested through clinics participating in the state's Infertility Prevention Project (IPP) and the incidence of gonorrhea among women as determined through public health reporting.

ELIGIBILITY:
With reference to the above question about sampling, we will measure PDPT use in a probability sample of persons with STD. Chlamydial prevalence will be measured in a sentinel population. Gonorrhea incidence will be based on public health surveillance.

Inclusion Criteria:

* All non-MSM with gonorrhea or chlamydial infection will be eligible for the study intervention.

Exclusion Criteria:

* MSM

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 33222 (Actual)
Dates: Start 2007-07; Primary Completion 2010-12 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Test positivity for Chlamydia trachomatis among women age 15-25 | October 2006 - December 2010
  The proportion of women age 15-25 testing positive for C. trachomatis in clinics participating in the WA State Infertility Prevention Project (IPP). Outcomes will be ascertained during five specified 3 month time periods occuring prior to the initiation of the study intervention in the four successive study waves and at the end of the study.
Gonorrhea incidence in women | October 2007-December 2010
  The incidence of gonorrhea in women in WA state local health jurisdictions as ascertained through public health reporting. Outcomes will be ascertained during five specified 3 month time periods occuring prior to the initiation of the study intervention in the four successive study waves and at the end of the study.

SECONDARY OUTCOMES:
Rates of recurrent gonorrhea | October 2007-Dec 2010
  Proportion of men and women with a second episode of gonorrhea occuring within 6 months of their initial diagnosis as ascertained through public health surveillance
Recurrent chlamydial infection | October 2006 - December 2010
  Proportion of men and women with a second episode of chlamydial infection occuring within 6 months of their initial diagnosis as ascertained through public health surveillance
Reported adverse drug reactions | July 2007-December 2010
  Adverse drug reactions reported to study staff following ingestion of medication supplied at patient delivered partner therapy. Outcome ascertained through passive surveillance.
Use of patient delivered partner therapy (PDPT) by medical providers | July 2007 - December 2010
  Proportion of persons with gonorrhea or chlamydial infection receiving PDPT from their diagnosing medical provider, excluding men who have sex with men

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Golden, MD, Principal Investigator — University of Washington
Locations (2):
- United States (2):
  - Washington State Department of Health, Olympia, Washington
  - University of Washington, Seattle, Washington

REFERENCES:
- [Background] Golden MR, Hughes JP, Brewer DD, Holmes KK, Whittington WL, Hogben M, Malinski C, Golding A, Handsfield HH. Evaluation of a population-based program of expedited partner therapy for gonorrhea and chlamydial infection. Sex Transm Dis. 2007 Aug;34(8):598-603. doi: 10.1097/01.olq.0000258319.54316.06. PMID 17413683
- [Derived] Golden MR, Kerani RP, Stenger M, Hughes JP, Aubin M, Malinski C, Holmes KK. Uptake and population-level impact of expedited partner therapy (EPT) on Chlamydia trachomatis and Neisseria gonorrhoeae: the Washington State community-level randomized trial of EPT. PLoS Med. 2015 Jan 15;12(1):e1001777. doi: 10.1371/journal.pmed.1001777. eCollection 2015 Jan. PMID 25590331